CLINICAL TRIAL: NCT07160829
Title: Focus on Levels of Awareness and Perceptions Regarding hsCRP in Identifying Systemic Inflammation in ASCVD, CKD and Heart Failure Management
Acronym: FLARE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-8416; U1111-1315-0755 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Atherosclerotic Cardiovascular Disease; Heart Failure; Chronic Kidney Disease
MeSH Terms: conditions — Atherosclerosis; Heart Failure; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nephrologist Group: This group includes nephrologists treating people with ASCVD and CKD.
  Interventions: Other: No treatment given
- Cardiologist Group: This group includes cardiologist treating people with ASCVD and CKD.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
This is a survey-based study conducted among cardiologists and nephrologists treating people with Atherosclerotic Cardiovascular Disease (ASCVD), Heart Failure (HF) and Chronic Kidney Disease (CKD). Study participants will be recruited to complete self-administered online survey. The purpose of this research is to gather real-world evidence related to attitudes around systemic inflammation and specifically the awareness, perception, drivers and barriers, and use of hsCRP in clinical practice to identify systemic inflammation in people with ASCVD+CKD and HF.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female, age above 18 years at the time of signing informed consent.
* Is a nephrologist or cardiologist. Cardiologists may be a mix of Interventional Cardiology, Heart Failure (HF) Specialist, General Cardiology, Preventative Cardiology, Cardiac Electrophysiology, Cardio-Oncology or Echocardiography (India only).
* Has been in specialty practice greater than or equal to 3 years.
* If cardiologist, sees at least 15 people with Atherosclerotic Cardiovascular Disease (ASCVD) with or without Chronic Kidney Disease (CKD) per month.
* If nephrologist, sees at least 20 people with ASCVD and CKD per month.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* If nephrologist, is only using dialysis to treat people with ASCVD and CKD.
* Does not meet inclusion criteria requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes cardiologists and nephrologists treating people with Atherosclerotic Cardiovascular Disease (ASCVD), Heart Failure (HF) and Chronic Kidney Disease (CKD)
Sampling Method: Non-Probability Sample
Enrollment: 608 (Actual)
Dates: Start 2025-09-18 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Perceptions towards role of systemic inflammation in identification, treatment, management of ASCVD+CKD and HF | At the time of survey response (Day 1)
  Multi-select from a defined list; 7-point Likert scale where 1=Not at all Important and Single-select from a defined list; Numerical; 7=Extremely Important; 7-point Likert scale where 1=Strongly Disagree and 7=Strongly Agree.
  Cardiologists and nephrologists' perceptions towards the role of systemic inflammation in the identification, treatment and management of people with Atherosclerotic Cardiovascular Disease and Chronic Kidney Disease (ASCVD+CKD) and Heart Failure (HF)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (4):
- Novo Nordisk Investigational Site, Sydney, Australia
- Novo Nordisk Investigational Site, Bangalore, Karnataka, India
- Novo Nordisk Investigational Site, Seoul, South Korea
- Novo Nordisk Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com